CLINICAL TRIAL: NCT02894255
Title: Prospective Multicenter Registry of Hybrid Coronary Artery Revascularization Combined With Surgical Bypass and Percutaneous Coronary Intervention Using Everolimus Eluting Metallic Stents
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Teikyo University (Other)
Responsible Party: Principal Investigator, Ken Kozuma, Professor, Teikyo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-233
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass; Percutaneous Coronary Intervention

ARMS (1):
- PCI and CABG (Experimental)
  Interventions: Device: Coronary artery bypass grafting; Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Device: Coronary artery bypass grafting
Procedure: Percutaneous coronary intervention

SUMMARY:
This prospective multicenter registry evaluates the efficacy of hybrid coronary revascularization (HCR) combining coronary artery bypass surgery (CABG) and percutaneous coronary intervention (PCI) in the treatment of multivessel coronary artery disease. CABG is to be performed in the left anterior descending artery and the left circumflex artery using only arterial grafts, whereas PCI is to be conducted for the treatment of significant stenotic disease in the right coronary artery with everolimus-eluting stents (EESs). This research plans to involve patients scheduled for coronary revascularization for multivessel coronary artery disease who consent to participate in the registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable angina, unstable angina, or non-ST elevation myocardial infarction.

  * Patients with multivessel coronary artery disease including significant stenotic lesion* in the right coronary artery and also including left main stem disease.
  * Patients who will be referred for CABG.
  * Patients with significant stenotic lesion in the right coronary artery amenable to PCI.
  * Patients who can take DAPT medications.
  * Patients who provided written informed consent. * Significant stenotic lesion means a condition where fractional flow reserve (FFR) is lower than 0.80 or visually confirmed stenosis is at least 75%.

Exclusion Criteria:

* • Patients with ST elevation myocardial infarction occurring within 24 hours before enrollment.

  * Patients who previously underwent CABG.
  * Patients who are at high risk of receiving CABG.
  * Patients who need simultaneous surgery such as valve surgery other than CABG.
  * Patients with a life expectancy of 1 year or shorter due to co-morbidities.
  * Patients with a history of cerebral infarction within the last 6 months.
  * Patients with congestive cardiac failure of NYHA 3 or higher.
  * Patients with unstable hemodynamics at enrollment.
  * Patients with right coronary artery disease that is chronic total occlusion and difficult to treat with PCI (J-CTO score of ≥ 23).
  * Patients receiving long-term dialysis.
  * Patients who are allergic to antiplatelet agent.
  * Patients who are critically allergic to contrast media.
  * Patients who are allergic to any DES component.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular event (death, myocardial infarction, cerebrovascular disorder, and repeat revascularization) | 12 months

REFERENCES:
- [Derived] Sugimoto K, Takahashi K, Okune M, Ueno M, Fujita T, Doi H, Tobaru T, Takanashi S, Kinoshita Y, Okawa Y, Fuku Y, Komiya T, Tsujita K, Fukui T, Shimokawa T, Watanabe Y, Kozuma K, Sakaguchi G, Nakazawa G. Impact of quantitative flow ratio on graft function in patients undergoing coronary artery bypass grafting. Cardiovasc Interv Ther. 2023 Oct;38(4):406-413. doi: 10.1007/s12928-023-00929-8. Epub 2023 Apr 5. PMID 37017900